CLINICAL TRIAL: NCT01770405
Title: Registry Trial for Clinical Evaluation of nCLE in Masses and Cystic Tumors of the Pancreas, Lymph Nodes, Submucosal Lesions of the GI Tract
Brief Title: Clinical Registry of nCLE in Masses and Cystic Tumors of the Pancreas, Lymph Nodes, Submucosal Lesions of the GI Tract
Acronym: US-nCLE
Status: Completed | Type: Observational
Sponsor: Mauna Kea Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: MKT_2012_nCLE_03
Record Dates: First submitted 2013-01-10; First posted 2013-01-17 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cyst; Pancreatic Neoplasms; Pancreatic Adenoma; Pancreatic Cancer; Pancreatic Islet Cell Tumors; Lymph Node Mass; Lymphadenopathy; GIST
Keywords: endomicroscopy; needle-based; pancreatic; cyst; mass; EUSFNA
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Neoplasms; Pancreatic adenoma; Adenoma, Islet Cell; Lymphadenopathy; Cysts; Arachnodactyly | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pancreatic cysts: Patient indicated for a first endoscopic ultrasound fine needle aspiration (EUS-FNA) for a pancreatic cyst,
  Interventions: Device: Endoscopic ultrasound fine needle aspiration

INTERVENTIONS:
Device: Endoscopic ultrasound fine needle aspiration — Device: nCLE needle-based Confocal Laser Endomicroscopy
  Other Names: ultrasonographic endoscopy; EUS-guided FNA

SUMMARY:
This study focuses on four different lesions: pancreatic cysts, lymph nodes near the gastrointestinal tract, pancreatic masses and GIST tumors.

On one hand, the results obtained during previous studies are more advanced for the assessment of the diagnostic performance of Cellvizio needle-based Confocal Laser Endomicroscopy (nCLE) system for Pancreatic cysts. Safety and technical feasibility have already been performed, and an interpretation criteria classification exists. On the other hand, results for pancreatic masses, Lymph nodes and GIST are less developed.

the objectives of the study are to

* Assess the diagnostic performance of the Cellvizio needle-based Confocal Laser Endomicroscopy (nCLE) system in diagnosing masses and cystic tumors of the pancreas, lymph nodes, submucosal lesions of the GI tract
* Define/Validate descriptive criteria of nCLE sequences in masses and cystic tu-mors of the pancreas, lymph nodes, submucosal lesions of the GI tract

DETAILED DESCRIPTION:
The principle of needle-based Confocal Laser Endomicroscopy (nCLE) is to image organs within or adjacent to the GI or respiratory tracts by means of a miniprobe inserted through an endoscopic needle. The fundamental technology, as well as the principle of operation of nCLE, is substantially similar to pCLE.

endoscopic fine needles are used during EUS-FNA procedures to puncture solid organs such as the pancreas, in order to get tissue or fluid for diagnostic purposes. There are different calibers of endoscopic nee-dles used. The most commonly used calibers for EUS-FNA procedures are 22G, 19G, and 25G needles. The nCLE Confocal Miniprobe is compatible with the 19G-type needle only. It is expected to help to differentiate the different types of lesions, especially for cysts, leading to better patient management. Microscopic tissue information in real-time in vivo during an EUS-FNA procedure may allow better differentiation between mucinous and non-mucinous cysts for instance.

ELIGIBILITY:
Inclusion Criteria:

* - Male or female > 18 years of age
* Patient indicated for a first EUS-FNA for masses and cystic tumors of the pancreas, lymph nodes, submu-cosal lesions of the GI tract
* Patients who had previous non-diagnostic tissue sampling taken during a previous EUS-FNA for masses and cystic tumors of the pancreas, lymph nodes, submucosal lesions of the GI tract
* Patient with known masses and cystic tumors of the pancreas, lymph nodes, submucosal lesions of the GI tract
* For pancreatic cyst patient, suffering chronic calcifying pancreatitis
* For pancreatic mass patient, any size or location
* For lymph node patient, any node reachable with EUS-FNA
* Willing and able to comply with study procedures and provide written informed consent to participate in the registry

Exclusion Criteria:

* - Subjects for whom EUS-FNA procedures are contraindicated
* Known allergy to fluorescein contrast
* If female, breast feeding or pregnant based on a positive hCG serum or an in vitro diagnostic test result
* Subject with multiple cysts
* Cysts <20 mm in diameter
* Previous EUS-FNA procedure performed less than 3 months ago
* If several pancreatic masses, only one will be imaged during the nCLE procedure
* Lymph nodes <5 mm in diameter
* If several suspicious lymph nodes, only the most suspect will be imaged during the nCLE proce-dure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Referral patients with a clinical indication for masses and cystic tumors of the pancreas, lymph nodes, submucosal lesions of the GI tract coming in for first EUS-FNA procedure at referral institution will be approached for possible inclusion into this registry
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
performance evaluation | up to one year
  * Assess the diagnostic performance of the Cellvizio needle-based Confocal Laser Endomicroscopy (nCLE) system in diagnosing masses and cystic tumors of the pancreas, lymph nodes, submucosal lesions of the GI tract (accuracy evaluation)
  * Define/Validate descriptive criteria for nCLE sequences in the characterization of masses and cystic tumors of the pancreas, lymph nodes, submucosal lesions of the GI tract (image interpretation criteria definition

SECONDARY OUTCOMES:
Safety and feasibility evaluation | up to one month following the procedure
  * Evaluate the feasibility and safety of nCLE for the characterization of masses and cystic tumors of the pan-creas, lymph nodes, submucosal lesions of the GI tract (IE. number of patients with complications, number of adverse events)
  * Build an atlas of images of nCLE sequences of masses and cystic tumors of the pancreas, lymph nodes, submucosal lesions of the GI tract

CONTACTS AND LOCATIONS:
Overall Officials: Divyesh V Sejpal, MD, Principal Investigator — Northwell Health
Locations (4):
- United States (4):
  - Emory University Hospital, Atlanta, Georgia
  - North Shore-LIJ Health System, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - Temple University Hospital, Philadelphia, Pennsylvania